CLINICAL TRIAL: NCT00597324
Title: Should Intervention Through RADial Approach be Denied to Patients With Negative Allen's Test Results?
Brief Title: Predictive Value of Allen's Test Result in Elective Patients Undergoing Coronary Catheterization Through Radial Approach
Acronym: RADAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marco Valgimigli (Other)
Responsible Party: Sponsor-Investigator, Marco Valgimigli, Head of the Catheterization laboratory, Università degli Studi di Ferrara
Organization: Università degli Studi di Ferrara (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-1-MV
Record Dates: First submitted 2007-12-26; First posted 2008-01-18 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Allen's test; lactate; safety; radial intervention; Patients with coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Patients with normal Allen's test
  Interventions: Procedure: coronary catheterisation
- 2 (Experimental): Patients with intermediate Allen's test
  Interventions: Procedure: coronary catheterisation
- 3 (Experimental): Patients with abnormal Allen's test
  Interventions: Procedure: coronary catheterisation

INTERVENTIONS:
Procedure: coronary catheterisation — Coronary angiography which may be followed by ad hoc percutaneous intervention if indicated clinically
  Other Names: Coronary angiography; PCI

SUMMARY:
The study will evaluate the feasibility and safety of radial approach in patients undergoing coronary catheterisation without any restrictions based on the results of Allen's test.

DETAILED DESCRIPTION:
The transfemoral access (TFA), through the percutaneous Seldinger technique, is the preferred approach in most catheterization laboratories worldwide due to its long history of use, the large availability of several dedicated preformed Judkins-type catheters and the possibility to exploit relatively large diameter catheters and sheaths, should these be necessary for complex percutaneous coronary intervention (PCI). Being a relatively deep and terminal vessel however, the femoral artery as percutaneous access site may expose to rare ischemic but frequent bleeding complications which occurs between 3-7% of patients undergoing interventional procedures, especially with modern anti-thrombotic drugs, including glycoprotein IIb/IIIa receptor blockers and clopidogrel. The difficulties in obtaining a stable and definitive local haemostasis, even when dedicated arterial vascular closure devices (VCD) are employed, make prolonged bed rest after TFA necessary in the majority of cases which result in patient discomfort and overall increase in medical expenditure.

In the last fifteen years, after Campeau's report of successful coronary angiography by transradial approach (TRA), the radial artery has been increasingly employed as an alternative access site both for diagnostic and interventional procedures.

The main advantage offered by percutaneous TRA is represented by the very low incidence of relevant vascular access site complications and bleeding and allows for early mobilization of the patient and thus to early discharge. As bleeding complications are increasingly recognized as strong and independent predictors of short and long-term outcomes following PCI, TRA may be the preferred access site by experienced teams. Radial artery (RA) cannulation, however, carries a risk of RA occlusion with an incidence of 4.8% to 19%. This is usually of no consequence, because the hand receives blood from both the radial and ulnar arteries (UA) with extensive collateral channels; however, some patients have incomplete palmar arches and might not have adequate communications between the ulnar and radial arteries. In these patients, there is a potential risk of hand ischemia in the event of RA occlusion.

A simple bedside test to check for communications between the ulnar and radial arteries is the modified Allen's test (AT). Patients with an abnormal test will usually have their cardiac catheterization performed via the femoral artery, thus denying them the potential advantages of transradial cardiac catheterization. In patients undergoing coronary angiography, the incidence of an abnormal AT ranges from 6.4% to 27%. Whether the AT can predict ischemic complications after RA cannulation is controversial, and some centers no longer exclude patients with an abnormal AT.

However, In 50 patients undergoing coronary angiography were screened for AT time. Circulation in the RA, UA, principal artery of the thumb (PAT), and thumb capillary lactate were measured before and after 30 min of RA occlusion. patients with an abnormal AT showed significantly reduced blood flow to the thumb and increased thumb capillary lactate (compared with patients with a normal AT) suggestive of ischemia. Based on these findings, Authors concluded that Transradial cardiac catheterization should not be performed in patients with an abnormal AT.

Aim of the RADAR study is to evaluate whether results of Allen's test in consecutive patients undergoing transradial coronary catheterization predict the occurrence of ischemic complications defined primarily as an increase of thumb capillary lactate and secondarily as a composite of local discomfort during and/or after the procedure, disability of the instrumented arm defined as perceived (subjective) or objective muscular weakness, need for surgical intervention or RA occlusion at any time within 30 days after catheterisation. Bleeding complications will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing coronary catheterisation through radial artery

Exclusion Criteria:

* Presence of haemodynamic instability
* Planned IABP insertion
* Previous trauma or surgical intervention in the instrumented arm
* Impossibility to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
elevation of thumb capillary lactate after the procedure | 30 days

SECONDARY OUTCOMES:
local discomfort, disability of the instrumented arm defined as perceived (subjective) or objective muscular weakness, need for surgical intervention or RA occlusion at any time within 30 days after catheterisation. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, PhD, Principal Investigator — Azienda Universitaria Ospedaliera di Ferrara, corso Giovecca 203; 44100; Ferrara; Italy
Locations (1):
- University Hospital, Ferrara, FE, Italy

REFERENCES:
- [Derived] Valgimigli M, Campo G, Penzo C, Tebaldi M, Biscaglia S, Ferrari R; RADAR Investigators. Transradial coronary catheterization and intervention across the whole spectrum of Allen test results. J Am Coll Cardiol. 2014 May 13;63(18):1833-41. doi: 10.1016/j.jacc.2013.12.043. Epub 2014 Feb 26. PMID 24583305